CLINICAL TRIAL: NCT00570388
Title: Neurocognitive Functioning Following The PROMETA® Treatment Protocol In Subjects With Alcohol Dependence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Addiction Medicine (Other)
Responsible Party: Jenny Starosta, Ph.D. and Joseph Volpicelli, MD, PhD- Co-Principal Investigator, Institute of Addiction Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20062166; WIRB Protocol Number: 20062166; WIRB Study Number: 1085483; WIRB Invest. Number: 128549
Record Dates: First submitted 2007-12-06; First posted 2007-12-10 (Estimated); Last update posted 2008-01-16 (Estimated); Status verified 2008-01

CONDITIONS: Alcohol Dependence
Keywords: Neurocognitive; Alcohol Dependence; Prometa; Prometa Protocol; Starosta
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Active Comparator): Subjects in the active Prometa group will receive flumazenil, gabapentin, and hydroxyzine per the Prometa Protocol.
  Interventions: Drug: Prometa Treatment Program
- 1 (Placebo Comparator): Subjects in the "placebo group" will receive placebo flumazenil, gabapentin, and hydroxyzine
  Interventions: Drug: Prometa Treatment Program

INTERVENTIONS:
Drug: Prometa Treatment Program — Day 1-3•Hydroxyzine HCL 50 mg and multivitamins with minerals po one hour before flumazenil infusion. Flumazenil infusion.
  Day 1•Gabapentin 300 mg po 9PM w/ hydroxyzine HCL 50 mg PRN for sleep.
  Day 2•Gabapentin 600 mg po 9PM w/ hydroxyzine HCL 50 mg PRN
  Day 3•Gabapentin 900 mg po 9PM w/ hydroxyzine HCL 50 mg PRN
  Days 4 through 28•Gabapentin 1200 mg po 9 PM
  Days 29 through 31•Gabapentin 900 mg po 9 PM
  Days 32 through 34•Gabapentin 600 mg po 9 PM
  Days 35 through 38•Gabapentin 300 mg po 9 PM
  Flumazenil Dosing Schedule
  2 mg flumazenil is given as a slow IV push. Subjects in the "placebo group" will receive placebo flumazenil, gabapentin, and hydroxyzine; subjects in the active group will receive flumazenil, gabapentin, and hydroxyzine per protocol.

SUMMARY:
This study will test the safety and efficacy of the PROMETA® Treatment Protocol (which includes the benzodiazepine antagonist flumazenil) in reversing the neurocognitive impairment and this in turn will lead to improved ability to resist alcohol related cues and enhance involvement in psychosocial treatment.

DETAILED DESCRIPTION:
The principal aim of this study is to extend our evaluation of the PROMETA® Treatment Protocol as a means to improve neurocognitive functioning in recently detoxified alcohol dependent subjects. For many alcohol dependent patients entering treatment, a range of neurocognitive deficits are present that not only had adverse effects on the patient's ability to function and think clearly but these deficits also impair the process of addiction treatment. For example, alcohol dependent subjects typically experience high levels of alcohol craving in the early stages of treatment. The patient is left with the choice of relieving craving by drinking alcohol to provide immediate relief of craving symptoms or abstaining from alcohol to obtain long-term benefits from recovery of the complications from excessive drinking. We have previously shown in open label trials that the PROMETA® Treatment Protocol helps stimulant abusers in the early stages of recovery, have relatively low rates of relapse to stimulant use. It is not clear if the Protocol is effective because of less urges to use stimulants or the ability to resist these urges is improved from a recovery of Neurocognitive functioning. The present proposal extends our previous research by comparing the efficacy of the PROMETA® Treatment Protocol in a double blind placebo controlled trial using a new population of substance abusers (alcohol dependent subjects) and assessing the effects of the PROMETA® Treatment Protocol on neurocognitive functioning, particularly those aspects of functioning that affect the ability to make decisions that have important long-term benefits.

ELIGIBILITY:
Inclusion Criteria:

* Patient must meet DSM-IV criteria for current diagnosis of alcohol dependence.
* In the past 30 days, patient had an average of >15 standard alcohol drinks/week with at least one day of five or more drinks.
* Patient must have successfully completed detoxification from alcohol (abstinent for three consecutive days). As evidenced by self-report or three negative breathalyzer reading and a CIWA-Ar score less than 6.
* Patient understands and signs the consent.

Exclusion Criteria:

* Patients with a current DSM-IV diagnosis of any substance dependence other than alcohol, nicotine, or cannabis.
* Patients with a current or past history of DSM-IV diagnosis of Panic Disorder
* Evidence of benzodiazepine use in the past 15 days, determined by self-report and/or by a urine drug screen
* Patients with a seizure disorder being managed with a benzodiazepine or for whom a benzodiazepine is being considered
* Patients who are currently being treated with psychotropic medications, including disulfiram, naltrexone, or acamprosate at the time of study entry.
* Patients with a history of unstable or serious medical illness, including need for benzodiazepines.
* Known severe physical or medical illnesses such as AIDS, active hepatitis,
* Current severe psychiatric symptoms, e.g., psychosis, dementia, acute suicidal or homicidal ideation, mania or depression requiring newly initiated antidepressant or psychotropic therapy, or which would make it unsafe for the patient to participate in the opinion of the primary investigator.
* Patients who have used investigational medication in the past 30 days.
* Female patients who are pregnant, nursing, or not using a reliable method of contraception.
* Patients with a condition that would make intravenous administration of medications difficult (e.g. absence of suitable peripheral veins).
* Have a known or hypersensitivity to medication components of PROMETA®TM
* Have been treated with PROMETA® for any reason currently or in the past year

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2007-03; Study Completion 2008-09 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure is neurocognitive functioning as assessed by a battery of standardized neurocognitive tests that assess, executive functioning, verbal memory, general intelligence, and attention. | Time Frame: Eight Weeks

SECONDARY OUTCOMES:
Secondary outcome measures include, alcohol craving, subject retention, percent of abstinent days, percent of heavy drinking days, time to first heavy drinking day, and blood chemistries including liver enzymes, reports of side effects. | Eight Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jenny J Starosta, PhD, Principal Investigator — Institute of Addiction Medicine; Joseph Volpicelli, MD, PhD, Principal Investigator — Institute of Addiction Medicine
Locations (1):
- Institute of Addiction Medicine, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Matching alcoholism treatments to client heterogeneity: treatment main effects and matching effects on drinking during treatment. Project MATCH Research Group. J Stud Alcohol. 1998 Nov;59(6):631-9. doi: 10.15288/jsa.1998.59.631. PMID 9811084
- [Background] Barker MJ, Greenwood KM, Jackson M, Crowe SF. Cognitive effects of long-term benzodiazepine use: a meta-analysis. CNS Drugs. 2004;18(1):37-48. doi: 10.2165/00023210-200418010-00004. PMID 14731058
- [Background] Bates ME, Pawlak AP, Tonigan JS, Buckman JF. Cognitive impairment influences drinking outcome by altering therapeutic mechanisms of change. Psychol Addict Behav. 2006 Sep;20(3):241-53. doi: 10.1037/0893-164X.20.3.241. PMID 16938062
- [Background] Girdler NM, Lyne JP, Wallace R, Neave N, Scholey A, Wesnes KA, Herman C. A randomised, controlled trial of cognitive and psychomotor recovery from midazolam sedation following reversal with oral flumazenil. Anaesthesia. 2002 Sep;57(9):868-76. doi: 10.1046/j.1365-2044.2002.02785.x. PMID 12190751
- [Background] Mason BJ. Treatment of alcohol-dependent outpatients with acamprosate: a clinical review. J Clin Psychiatry. 2001;62 Suppl 20:42-8. PMID 11584875
- [Background] Mason BJ, Goodman AM, Chabac S, Lehert P. Effect of oral acamprosate on abstinence in patients with alcohol dependence in a double-blind, placebo-controlled trial: the role of patient motivation. J Psychiatr Res. 2006 Aug;40(5):383-93. doi: 10.1016/j.jpsychires.2006.02.002. Epub 2006 Mar 20. PMID 16546214
- [Background] Rupp CI, Fleischhacker WW, Drexler A, Hausmann A, Hinterhuber H, Kurz M. Executive function and memory in relation to olfactory deficits in alcohol-dependent patients. Alcohol Clin Exp Res. 2006 Aug;30(8):1355-62. doi: 10.1111/j.1530-0277.2006.00162.x. PMID 16899038
- [Background] Singh N, Sharma A, Singh M. Possible mechanism of alprazolam-induced amnesia in mice. Pharmacology. 1998 Jan;56(1):46-50. doi: 10.1159/000028181. PMID 9467187
- [Background] Srisurapanont M, Jarusuraisin N. Opioid antagonists for alcohol dependence. Cochrane Database Syst Rev. 2005 Jan 25;(1):CD001867. doi: 10.1002/14651858.CD001867.pub2. PMID 15674887
- [Background] Stewart SA. The effects of benzodiazepines on cognition. J Clin Psychiatry. 2005;66 Suppl 2:9-13. PMID 15762814
- [Background] Tapert SF, Ozyurt SS, Myers MG, Brown SA. Neurocognitive ability in adults coping with alcohol and drug relapse temptations. Am J Drug Alcohol Abuse. 2004 May;30(2):445-60. doi: 10.1081/ada-120037387. PMID 15230085
- [Background] Uekermann J, Daum I, Schlebusch P, Wiebel B, Trenckmann U. Depression and cognitive functioning in alcoholism. Addiction. 2003 Nov;98(11):1521-9. doi: 10.1046/j.1360-0443.2003.00526.x. PMID 14616178
- [Background] Zinn S, Stein R, Swartzwelder HS. Executive functioning early in abstinence from alcohol. Alcohol Clin Exp Res. 2004 Sep;28(9):1338-46. doi: 10.1097/01.alc.0000139814.81811.62. PMID 15365304